CLINICAL TRIAL: NCT05535114
Title: The Effects of an Intradialytic Yoga-Resistance Exercise on Muscle Strength, Fatigue, Depression, and Sleep Quality in Hemodialysis Patients: a Randomized Controlled Trial
Brief Title: Intradialytic Yoga-resistance Exercise for Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Bach Mai Hospital (Other)
Responsible Party: Principal Investigator, Tsae Jyy, Wang, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2431/BM-HĐĐĐ
Record Dates: First submitted 2022-08-30; First posted 2022-09-10 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-07

CONDITIONS: Hemodialysis
Keywords: intra-dialytic yoga-resistance exercise; hemodialysis; muscle strength; fatigue; sleep quality; depression; body composition
MeSH Terms: conditions — Fatigue; Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga-resistance exercise (YRE) group (Experimental): The YRE group will perform breathing exercises, flexibility, resistance exercises and relaxation. It will be carried out for about 30 to 45 minutes in the first two hours of each hemodialysis session, three times weekly for 12 weeks. The intensity of resistance exercise will be adjusted individually at week 3, week 7, and week 11 to the rate of perceived exertion of "somewhat hard" (on the Borg scale 6-20). The intensity of resistance exercise will be increased gradually by changing the different colors of elastic bands.
  Interventions: Other: Yoga-resistance exercise
- Control group (No Intervention): Participants in the control group will receive only usual care. They will be able to receive the YRE protocol after completing the study.

INTERVENTIONS:
Other: Yoga-resistance exercise — Breathing exercise (5 minutes), flexibility (5 minutes), resistance exercise (20 minutes), relaxation & meditation (10 minutes).
  Arms: Yoga-resistance exercise (YRE) group

SUMMARY:
Objective: Intra-dialytic exercises are strongly believed to have benefits and have become a crucial therapeutic modality for managing hemodialysis patients. The effects of each type of exercise and yoga on hemodialysis patients' physical and psychological health have been studied extensively. However, the effects of combining yoga and resistance training exercises remain unclear in this population. The aims of this study are: (1) to create a feasible intradialytic yoga-resistance exercise (YRE) program for hemodialysis patients; and (2) to investigate its effects on muscle strength, fatigue, depression, and sleep quality in hemodialysis patients.

Methods: Seventy-two participants will be randomly assigned to a 12-week YRE group or a wait-list control group. The YRE group will perform exercises (breathing exercises, flexibility, resistance exercises, relaxation with meditation) in the first two hours of each hemodialysis session, three times weekly. The outcome measures are the following: socio-demographic characteristics; fatigue (measured by the Functional Assessment of Chronic Illness Therapy-Fatigue); depression (the Patient Health Questionnaire); sleep quality (Pittsburgh Sleep Quality Index); muscle strength (a hydraulic hand dynamometer, hand-held dynamometer, and one-minute sit-to-stand test). The outcomes will be assessed at baseline, week 6, and week 12. The independent t-test will be applied to compare the differences in outcome scores between groups at different time points. Using a generalized estimating equation method to analyze the effects of the intervention on the outcome variables.

Results: The expected results are: (1) The combined YRE program is feasible and safe for hemodialysis patients. (2) After 12 weeks, the intervention group will show significant improvement in muscle strength, fatigue, depression, and sleep quality compared to the control group.

DETAILED DESCRIPTION:
Study design: a randomized controlled trial.

Setting: This study will be conducted at the dialysis department of the Bach Mai hospital which is a national-level hospital in Hanoi, Vietnam.

Sample size: The sample size was calculated using G*Power software 3.1.9.7 (Faul et al., 2007) with α = 0.05, the 1-beta error probability of 0.80, and the effect size for the main outcome of the leg muscle strength was 0.66 (Rosa et al., 2018). A sample size of 30 participants for each group was calculated. Anticipating a 20% attrition rate, a total number of 36 participants is assigned to each group.

Recruitment process: The potentially eligible participants will be referred by the head nurse or the nephrologists at the Dialysis Department of Bach Mai hospital. The researcher will assess the potential participants' eligibility via their medical records and cognitive and physical function assessment as well as reconfirm with their nephrologists. The researcher will explain the study's purpose, procedures, potential benefits, and risks of participating in this study to patients and their families.

Randomization & allocation concealment: The randomization procedure will be performed by a nurse lecturer who does not participate in the study recruitment and data collection.

To prevent intervention diffusion, the participants will be randomly assigned to the intervention group or the control group according to their hemodialysis (HD) schedules.

Intervention: The protocol of the combined YRE program will be generated based on findings obtained from a literature review. It consists of four parts as follows: breathing exercises, flexibility, strength exercises and relaxation. It will be carried out about 30 minutes to 45 minutes in the first two hours of each HD session after connecting the patient to the dialysis machine for 30 minutes, three times weekly for 12 weeks.

Due to the facility conditions and fall prevention purposes, all types of exercise in the combined YRE program will be done when in the supine position.

The intensity of the resistance training: During the first two weeks of training, the participants will perform two sets of 8-12 repetitions for each type of strength exercise with the yellow or red elastic band depending on the participant's tolerance. Three sets of each exercise will apply from the third week until the end. The rest interval between sets and exercises is one to two minutes. The training intensity will be adjusted at week 3, week 7, and week 11 according to the increase in muscle strength. The intensity of each strength exercise will be increased gradually by changing the different colors of elastic bands. The intensity of strength exercise that each patient can tolerate will be adjusted to the rate of perceived exertion (RPE) of "somewhat hard" (13-14 on the Borg scale) (Borg, 1982).

Validation of the combined YRE program: This protocol will be validated the suitability by a panel of experts before implementing in the feasibility study. The experts include one physiotherapist; one nephrologist, one hemodialysis nurse, and one yoga teacher.

Interventionist: the researcher and another HD nurse (at least five years' experiences experience in working with HD patients).

Intervention delivering: A pre-training information session will be given to all participants one week before the intervention at the dialysis unit by the interventionists. The first two weeks, participants will be familiarized with the intervention. In the following weeks, the participants will practice exercises under the interventionist's supervision.

Monitor for safety, adverse events: All potentially eligible participants will be confirmed by their nephrologists for exercise capacity before recruiting for this study. The blood pressure, heart rate, and SpO2 will be monitored before and after training. The interventionists will supervise the patient's exercise and monitor for exercise-related side effects such as nausea or vomiting; a sudden headache, dizziness, or a feeling of lightheadedness; a sudden weakness in your arms or legs; hypotension. Stop exercise and medical consultation will be recommended if any of these problems occur. Moreover, other side-effects of exercise such as muscle soreness, joint problems, or injuries should also be documented.

Data collection: Data collection will be done at the baseline, week 6, and week 12 on a midweek non-dialysis day. The data collector (A nephrology nurse) will be blinded to the study group assignment. It takes about 30 minutes.

Feasibility & Safe of the YRE: The feasibility of the recruitment process, The attrition rate The adherence rate, Length of time for intervention implementation, Adverse events associated with the intervention.

Instruments The study questionnaires include questions on demographics (age, gender, marital status, education, occupation), The Functional Assessment of Cancer Therapy-Fatigue (FACIT-F), Patient Health Questionnaire (PHQ-9), and sleep quality (Pittsburgh Sleep Quality Index). Disease characteristics, including body height (cm), weight after dialysis (kg), body mass index (BMI, kg/m2), HD vintage (years), HD access site, and Charlson comorbidity index will be collected from the participants' medical records. The physical measurements include muscle strength measures of upper limbs and lower limbs, and one-minute STS test.

Data analysis: Using independent t-test and chi-square tests to test the homogeneity of two groups at baseline. The independent t-test will be applied to compare the differences on outcome's scores between groups in different time points. A generalized estimating equations method will be used to analyze the effect of the intervention on the outcome variables.

Ethical consideration: Ethical approvals will be obtained from the Ethical Committee of Hanoi Medical University, Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ESRD
* Undergoing maintenance hemodialysis treatment for more than three months,
* Age between 45 years and 65 years old,
* Under the permission of their nephrologist,
* Able to communicate in Vietnamese.

Exclusion Criteria:

* Unstable cardiac status such as angina, heart failure stage ≥ 3, myocardial infarction in the last six months, uncontrolled arrhythmia, uncontrolled hypertension with systolic blood pressure ≥ 200 mmHg or diastolic blood pressure ≥ 120 mmHg, symptomatic tachyarrhythmia or bradyarrhythmias, cardiovascular stent implantation, pacemaker installation,
* Artificial joint replacement; amputations or prostheses in upper and lower extremities,
* Suspected or known dissecting aneurysm,
* Uncontrolled diabetes (blood sugar 2 hours after eating < 7 or > 14 mmol),
* Hospitalization during the previous month, except for vascular access repair,
* Currently or in previous month (≥ three times/week) involved in any exercise program (e.g. yoga, aerobic, taichi…),
* Arteriovenous fistula dysfunction or new central venous catheter/ arteriovenous fistula access (less than 3 months)
* Severe cognitive impairment (screened by the nephrologist)
* Currently taking an antidepressant

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Muscle strength- "change" is being assessed | Pre-test (before intervention start); Post-test one (at week 6); Post-test two (at week 12)
  Handgrip strength will be measured by a dynamometer (NY 10602 USA). The test-retest reliability of this equipment was confirmed in a previous study (Savva et al., 2014).
  Extension/flexion of elbow, shoulder, and hip; and hip abduction/adduction will be assessed by the handheld dynamometer (USA, model 01163). Validity and reliability of a handheld dynamometer in measuring upper limb strength have been confirmed (Chen et al., 2021). We use the testing protocol reported from a prior study (Andrews et al., 1996).
  One-minute STS test: It is a valid and reliable measures of lower limb muscle strength (Segura-Ortí & Martínez-Olmos, 2011). The number of repetitions of sitting down and getting up from a chair in one minute will be recorded.

SECONDARY OUTCOMES:
The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Pre-test (before intervention start); Post-test one (at week 6); Post-test two (at week 12)
  The FACIT-F, a subscale of the FACIT tool, will be used to assess the level of fatigue and its impact on daily activities and function over the previous seven days (Yellen et al., 1997). It is short and easy to administer, which consists of 13 items graded on a five-point Likert scale (0 = not at all fatigued; 1 = a little bit fatigued; 2 = somewhat fatigued; 3 = quite a bit fatigued; and 4 = very much fatigued). The total score ranges from 0 to 52. High scores represent more fatigue. The FACIT-F has showed as a reliable and valid instrument (Long et al., 2016; Wang et al., 2015). This instrument has been also used in hemodialysis patients and in Vietnamese population. It will be used three times to see how yoga-resistance exercise will change fatigue level in hemodialysis patients before and after intervention.
Patient Health Questionnaire (PHQ-9) | Pre-test (before intervention start); Post-test one (at week 6); Post-test two (at week 12)
  The PHQ-9 will be used to measure participants' depression severity (Kroenke et al., 2001). It is a valid and reliable tool for using in the hemodialysis population (Alshraifeen et al., 2020; Thomas et al., 2017). High internal consistency and test-retest reliability has been demonstrated in previous studies (Kroenke et al., 2001; Nguyen et al., 2022). The tool was also validated and used in Vietnamese population (Dang et al., 2022; Nguyen et al., 2022). There are nine items in the scale indicating nine depressive symptoms. Patients will be asked to self-report each depressive symptom that they have experienced over the last two weeks on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). The total score of the nine items represent the scale score, with a possible range of 0 to 27. A score of 10 or above is classified as depression (Kroenke et al., 2001).
The Pittsburgh Sleep Quality Index (PSQI)- "change" is being assessed | Pre-test (before intervention start); Post-test one (at week 6); Post-test two (at week 12)
  Using PSQI to measure sleep quality (Buysse et al., 1989). It has been widely used in hemodialysis population. It has also been validated and used in the Vietnamese population (Nguyen et al., 2018). The reliability and validity of this scale have been confirmed in previous studies (Maniam et al., 2014). It consists 19 self-reported questions to assess sleep quality, frequency and severity of specific sleep-related problems during the prior month. There are seven domains including sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medications and daytime dysfunctions. Each component score is calculated and coded from 0 to 3 (0 = very good; 1 = fairly good; 2 = fairly bad; 3 = very bad). The total score of PSQI ranges from 0 to 21, with a higher score indicating lower sleep quality.
Body composition | Pre-test (before intervention start); Post-test one (at week 6); Post-test two (at week 12)
  Body composition includes body height (m), weight after dialysis (kg), body mass index (BMI, kg/m2), body mass (Kg), Body fat ratio (%), Visceral fat level (0.5 level), Protein (kg) will be measured by Using Health-care Box (HcBox). HcBox is a mobile health monitoring system supported by the AI365 (Artificial Intelligence Health Advice Push System), CRM (Customer Relationship Management) system, and WowGoHealth APP.
International Physical Activity Questionnaire short version (IPAQ-SF) | Pre-test (before intervention start); Post-test one (at week 6); Post-test two (at week 12)
  We will use the IPAQ-SF (Craig et al., 2003) to assess physical activity level which will be treated as covariate of outcomes. Patients will be asked to provide information about their time spent on sitting, walking, moderate and vigorous physical activities during the last seven days. The IPAQ was used in the Vietnamese population (Nguyen & Do, 2021). The overall physical activity score is calculated by multiplying minutes spent on activities at different levels including sitting, walking, moderate, and vigorous, by 1.0, 3.3, 4.0, and 8.0, respectively (Craig et al., 2003; Nguyen & Do, 2021). The metabolic equivalent task scored in minutes per week (MET-min/wk) was used as the measuring unit of physical activity (Lee et al., 2011).
The 5-item healthy eating score (HSE) | Pre-test (before intervention start); Post-test one (at week 6); Post-test two (at week 12)
  Using the 5-item HSE (Purvis et al., 2013; Shams-White et al., 2019) to assess dietary intake behavior which will be treated as covariate. This tool was used in Vietnamese population (Vu et al., 2021). Hemodialysis patients will report their frequency consumption of fruits, vegetables, whole grains, dairy, and fish over the last 30 days on a five-point scale with 0 being "rarely or never", 1 being "1-2 times/week", 2 being "3-6 times/week", 3 being "once/day", 4 being "twice/day", and 5 being "3 or more times/day". The total HES scores range from 0 to 25, the higher score the better healthy eating behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Bach Mai Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://doi.org/10.1007/s10943-020-00988-8
- See also: Related Info — https://doi.org/10.1016/0165-1781(89)90047-4
- See also: Related Info — https://doi.org/10.1123/jsr.2020-0021
- See also: Related Info — https://doi.org/10.1249/01.mss.0000078924.61453.fb
- See also: Related Info — https://doi.org/10.1046/j.1525-1497.2001.016009606.x
- See also: Related Info — https://doi.org/10.1186/1479-5868-8-115
- See also: Related Info — https://doi.org/10.1016/j.ejon.2015.10.010
- See also: Related Info — https://doi.org/10.11622/smedj.2014119
- See also: Related Info — https://doi.org/https://doi.org/10.1016/j.jpainsymman.2018.02.019
- See also: Related Info — https://doi.org/10.1007/978-3-030-75506-5_72
- See also: Related Info — https://doi.org/https://doi.org/10.1016/j.jmpt.2014.02.001
- See also: Related Info — https://doi.org/10.2215/cjn.03900417
- See also: Related Info — https://doi.org/10.1016/j.jpainsymman.2014.04.011
- See also: Related Info — https://doi.org/10.1016/s0885-3924(96)00274-6